CLINICAL TRIAL: NCT05966181
Title: The Effect of Repeated Simulation in Developing Social Justice Advocacy Attitudes and Skills on Nursing Student
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esin Ateş, research assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ege Uni-NF-11
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Nurse's Role; Education; Nursing
Keywords: Social justice; advocacy; repeated simulation

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study with pretest-posttest control group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): They will perform repetitive simulation (standard patient simulation according to scenarios) with the students in the experimental group.
  Interventions: Behavioral: experimental group
- control group (Other): A single simulation will be applied to the control group (standard patient simulation according to scenarios).
  Interventions: Behavioral: experimental group

INTERVENTIONS:
Behavioral: experimental group — Experimental Group-Repetitive Simulation
  * First simulation application; It will be done in groups of four with a total of 5 groups (n=20). In each scenario, one student in the group will participate in the role of nurse and three other students will participate as audience. Four students in each group will take part in a standard patient simulation consisting of four different scenarios.
  * Second simulation application; It will be carried out with the students in the experimental group about 3-4 weeks after the first simulation. Each student will use one new scenario alone in the second simulation.

SUMMARY:
It is a randomized controlled experimental and single-blind study with a pretest-posttest control group design.

DETAILED DESCRIPTION:
It is a randomized controlled experimental and single-blind study with a pretest-posttest control group design, planned to examine the effect of repeated simulation (standard patient simulation) on improving nursing students' social justice advocacy attitudes and skills.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research Being a 4th year undergraduate nursing student Having completed the theoretical education for vocational courses

Exclusion Criteria:

* Being a foreign national (due to Turkish speaking/understanding problem)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Repeated simulation | four weeks
  Repeated simulation is effective in developing nursing students' social justice advocacy attitudes and skills.
  Students' social justice advocacy attitudes will be measured with the "Social Justice Advocacy Scale". The scale is a 7-point Likert-type scale. 1 means "Absolutely Not True" and 7 means "Absolutely True". The minimum score is 41 and the maximum score is 287 from the scale; it is stated that as the scores obtained from the scale increase, social justice advocacy skills also increase.
  Students' advocacy skills will be measured with the "Social Justice Advocacy Skills Assessment Guide". The scoring in the guide was as follows: "Not Done = 0, insufficient performance = 1 and sufficient performance = 2.". The minimum score received from the guide is 0 and the maximum score is 48; as the total score received from the guide increases, the students' advocacy application skill levels are considered to be higher.

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Özsoy, Prof, Study Chair — suheyla.ozsoy@ege.edu.tr
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No